CLINICAL TRIAL: NCT05320614
Title: The Effect Of Web-Based Educatıon And Therapeutıc Game Method Gıven To Chıldren In Planned Surgery On Pre-Surgery Anxıety And Fear On Post-Operatıve Paın And Sleep
Brief Title: Education for Children Who Will Have Planned Surgery With Web-based and Therapeutic Game Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Collaborators: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Derya Demir Uysal, lecturer, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MSKU UYSAL-001
Record Dates: First submitted 2022-03-04; First posted 2022-04-11 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Day Surgery
Keywords: Web-based education,; therapeutic play; anxiety; pain; fear
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case 1 (Experimental): Case Group:Web-Based Education Information about the operation that the child will undergo; animation films about the hospital, the operating room and the medical equipment to be used; training with presentation including methods of coping with anxiety, fear and pain, postoperative wound care, possible complications in nutrition and nursing care; educational games Education with Therapeutic Play Method Training with the therapeutic game method for 30-45 minutes in the game room in the service one day before the surgery
  Interventions: Other: Web-Based Education
- control 1 (Experimental): Control Group: Explaining the routine care given in the service by the pediatric surgery nurse to the child and parent in the control group.
  Interventions: Other: Routine maintenance Training

INTERVENTIONS:
Other: Web-Based Education — Web-Based Education Information about the operation that the child will undergo; animation films about the hospital, the operating room and the medical equipment to be used; training with presentation including methods of coping with anxiety, fear and pain, postoperative wound care, possible complications in nutrition and nursing care; educational games Education with Therapeutic Play Method Training with the therapeutic game method for 30-45 minutes in the game room in the service one day before the surgery
  Arms: case 1
Other: Routine maintenance Training — Explaining the routine care given to the child and parent in the control group by the pediatric surgery nurse in the service.
  Arms: control 1

SUMMARY:
This research was planned to determine the effects of the web-based education given at home to children aged 7-12 in planned surgeries and the therapeutic game method applied in the hospital on pre-operative anxiety and fear, postoperative pain and sleep.

This study is a randomized controlled experimental study.

DETAILED DESCRIPTION:
Illness and especially hospitalization in the preoperative and postoperative period cause trauma with physiological, emotional and behavioral problems for children. With the help of web-based education and therapeutic game methods by pediatric nurses, anxiety, fear and pain seen in children and families can be reduced and skills to cope with negative emotions can be improved.

This research was planned to determine the effects of the web-based education given at home to children aged 7-12 in planned surgeries and the therapeutic game method applied in the hospital on pre-operative anxiety and fear, postoperative pain and sleep.

This study is a randomized controlled experimental study. The study is planned to be performed in the pediatric surgery clinic of the Training and Research Hospital.

For sample selection, children will be stratified in terms of age variables and divided into two strata as 7-9 years old and 10-12 years old. In order to ensure homogeneity between the groups, children will be selected into the study and control groups using a simple randomization method and a random numbers table. To the children in the study group and their parents; information about the child's surgery, educational brochures including the conditions to be considered before, during and after the operation, during the discharge period, operating room tour, educational games, etc. Training will be given on the website using and a therapeutic game will be played in the game room at the hospital the day before the surgery. The children in the control group and their parents will be given routine care and information about the pre-operative preparation in the service. Descriptive statistics, Chi-square test will be used in the evaluation of the data. A value of p<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* Those who will have a planned surgery between the ages of 7-12,
* Having and able to use a computer/tablet and internet connection at home,
* Having the ability to use a computer / tablet,
* Pediatric patients given written consent by their parents

Exclusion Criteria:

* At least one previous experience of surgery
* Having communication problems (sight, hearing, mental),
* Diagnosed with anxiety disorder,
* Genetic/congenital disease,

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Child Fear Scale: | On the day of the operation, one hour before the operation, the child is asked to rate his/her fear according to this scale.
  This scale is scored between 0-4 based on five different facial expressions, a higher scale score indicates more fear.

SECONDARY OUTCOMES:
Yale Modified Preoperative Anxiety Scale Child Form | An evaluation is made by the researcher 30 minutes before the operation and when the anesthesia mask is shown in the operating room.
  This scale has four parameters, each parameter is scored between 0-4, the second parameter is scored between 0-6. A total of minimum 4 and maximum 18 points can be obtained from the scale. High scores indicate high anxiety.

OTHER OUTCOMES:
Wong-Baker Facial Pain Scale | An evaluation is made by asking the child to rate his/her pain according to this scale, two hours after he/she comes to the service room after the surgery and before being discharged.
  This scale is used to determine the level of pain in children aged 3-18 years. There are six face shapes in the scale, and as you go from left to right, the expression of the faces worsens to show the severity of pain. Accordingly, the leftmost facial expression means "I feel good", and the rightmost facial expression means "I feel extremely bad". Evaluation of the scale is based on the principle of asking the child to mark the face shape that expresses his/her condition. Scoring is done as 0-10 points.
Sleep Disturbance Scale For Children | It is filled ten days after the operation. When the child comes to the check-up ten days after discharge from the hospital, the evaluation is completed by the parent in the polyclinic.
  It is a Likert-type scale that investigates sleep disorders in children aged 6-16 years that have occurred in the last six months. In the scale, the child's sleep disorders are questioned in 26 items and 6 sub-dimensions. Questions are answered from never (1 point) to always (5 points). A total of minimum 26 and maximum 130 points can be obtained from the scale. Higher scores indicate more sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Hüsniye ÇALIŞIR, Prof.Dr, Study Director — Aydin Adnan Menderes University
Locations (2):
- Turkey (Türkiye) (2):
  - MSKU, Muğla, Menteşe
  - Derya DEMİR UYSAL, Muğla

IPD SHARING:
Plan to Share IPD: No